CLINICAL TRIAL: NCT02411344
Title: PERtuzumab-trastuzumab Plus lEetrozoLe In Endocrine Sensitive Breast Cancer: a Phase II neoAdjuvant Study
Brief Title: Preoperative Study With Trastuzumab, Pertuzumab and Letrozole in Breast Cancer Patients Sensitive to Hormonal Therapy
Acronym: PER-ELISA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Oncologico Veneto IRCCS (Other)
Collaborators: Association for Translational Research in Oncology (AS.T.R.O.) (Unknown)
Responsible Party: Principal Investigator, Valentina Guarneri, MD, PhD, Istituto Oncologico Veneto IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AS.T.R.O.BC01-13; 2013-002662-40 (EudraCT Number)
Record Dates: First submitted 2015-03-05; First posted 2015-04-08 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Endocrine Sensitive HER2+/HR+ Breast Cancer
Keywords: HER2+/HR+; breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pertuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pertuzumab, Trastuzumab, Letrozole (Experimental)
  Interventions: Drug: Pertuzumab

INTERVENTIONS:
Drug: Pertuzumab — * Pertuzumab 840 mg loading dose iv on day one, followed by 420 mg iv every 3 weeks for 5 cycles
  * Trastuzumab 8 mg/kg loading dose iv on day 2, followed by 6 mg/kg iv on day 2 of each subsequent 3 weekly cycle
  * Letrozole 2.5 mg daily p.o. for five 21-day cycles (to be continued until surgery).
  Other Names: Perjeta

SUMMARY:
The purpose of this study is to evaluate the activity of molecular response in endocrine sensitive breast cancer HER2+/HR+ patients treated with Pertuzumab-trastuzumab plus Ietrozole.

DETAILED DESCRIPTION:
The purpose of this study is:

* to evaluate the rate of pathologic complete response (pCR), as defined as complete disappearance of invasive tumor in breast and axillary nodes.
* to estimate the percentage of clinical objective responses (cOR) (complete plus partial) in the breast, as assessed by ultrasonography (US)
* to estimate the percentage of breast conservative surgery
* to evaluate the safety profile
* To perform correlative biomarker analyses

ELIGIBILITY:
Inclusion Criteria:

* primary diagnosis of infiltrating breast cancer
* HR positivity (ER ≥ 10% and/or PgR ≥10%) and HER2 positivity (IHC 3+ or FISH/CISH amplification), as assessed by local laboratory.
* Stage II-IIIA
* age >18 yrs
* ECOG Performance Status 0-1
* Postmenopausal status, defined by at least one of the following:

  60 years of age; < 60 years of age and amenorrheic for >/=12 months prior to day 1 < 60 years of age, without a uterus, and luteinizing hormone (LH) and follicle stimulating hormone (FSH) values within postmenopausal range Prior bilateral oophorectomy Prior radiation castration with amenorrhea for at least 6 months
* Cardiac ejection fraction within the institutional range of normal (as measured by echocardiogram or MUGA scan).
* Normal organ and marrow function as defined below:

(leukocytes >=3000/mcL; absolute neutrophil count >=1,500/mcL; platelets >=100,000/mcL; total bilirubin within 1.25 x normal institutional limits (with the exception of Gilbert's syndrome); AST (SGOT)/ALT(SGPT) within 1.25 x institutional upper limit of normal creatinine within normal institutional limits

* Availability of tumor tissue suitable for biological and molecular examination before starting primary treatment
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Stage IIIB, IIIC, and inflammatory breast cancer
* Stage IV breast cancer
* Prior treatment with chemotherapy, endocrine therapy or radiotherapy. Prior treatment with HER2 targeting therapies
* LVEF below the ULN
* Uncontrolled hypertension (systolic >150 mm Hg and/or diastolic >100 mm Hg) or clinically significant (i.e. active) cardiovascular disease: cerebrovascular accident (CVA)/stroke or myocardial infarction within 6 months prior to first study medication, unstable angina, congestive heart failure (CHF) of New York Heart Association (NYHA) grade II or higher, or serious cardiac arrhythmia requiring medication.
* Received any investigational treatment within 4 weeks of study start.
* Subjects with known infection with HIV, HBV, HCV
* Known hypersensitivity to any of the study drugs or excipients.
* Dyspnoea at rest or other disease requiring continuous oxygen therapy.
* Psychiatric illness/social situations that would limit compliance with study requirements
* Subjects assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-02; Primary Completion 2018-01-12 (Actual); Study Completion 2018-01-12 (Actual)

PRIMARY OUTCOMES:
Rate of pathologic complete response | At time of surgery, within 3 weeks from the last i.v. therapy
  A pathologic complete response (pCR) is defined the complete absence of infiltrating tumor cells in the breast and in lymph nodes. Residual in situ disease (DCIS) will be included in the pCR category.

SECONDARY OUTCOMES:
Percentage of clinical objective response. | At time of surgery, within 3 weeks from the last i.v. therapy
  The Clinical Response will be defined according to RECIST criteria comparing the tumor size (largest tumor diameter) before and after treatment, as assessed by ultrasound examination.
Rate of Conservative Surgery | At time of surgery, within 3 weeks from the last i.v. therapy
Safety profile assessed by the NCI Common Terminology Criteria for Adverse Events (CTCAE) To version 4.0 will be used | Every 21-day cycles
Occurrence of mutations in the PIK3CA gene | Within 4 weeks prior to first dose treatment

CONTACTS AND LOCATIONS:
Overall Officials: Valentina Guarneri, MD; PhD, Principal Investigator — Medical Oncology 2, Istituto Oncologico Veneto
Locations (8):
- Italy (8):
  - Policlinico Vittorio Emanuele, Catania, CT
  - Arcispedale S. Anna, Cona, FE
  - Istituto Europeo di Oncologia, Milan, MI
  - Istituto Nazionale Tumori, Milan, MI
  - Ospedale "Guglielmo da Saliceto", Piacenza, PC
  - Istituto Oncologico Veneto, Oncologia Medica 2, Padua, PD
  - Arcispedale S. Maria Nuova, Reggio Emilia, RE
  - A. O. U. Santa Maria della Misericordia, Udine, UD

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guarneri V, Dieci MV, Bisagni G, Frassoldati A, Bianchi GV, De Salvo GL, Orvieto E, Urso L, Pascual T, Pare L, Galvan P, Ambroggi M, Giorgi CA, Moretti G, Griguolo G, Vicini R, Prat A, Conte PF. De-escalated therapy for HR+/HER2+ breast cancer patients with Ki67 response after 2-week letrozole: results of the PerELISA neoadjuvant study. Ann Oncol. 2019 Jun 1;30(6):921-926. doi: 10.1093/annonc/mdz055. PMID 30778520